CLINICAL TRIAL: NCT00133536
Title: A Randomized, Double-Blinded, Placebo-Controlled, Phase I/II, Study of the Safety, Reactogenicity, and Immunogenicity of Intramuscular Inactivated Influenza A/H5N1 Vaccine in Healthy Children Aged 2 Years Through 9 Years
Brief Title: A/H5N1 Vaccine in Healthy Children Aged 2-9 Years
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Robert Johnson, HHS/NIAID/DMID
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 04-077
Record Dates: First submitted 2005-08-19; First posted 2005-08-23 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2008-06

CONDITIONS: Influenza
Keywords: H5N1, Influenza, children
MeSH Terms: conditions — Influenza, Human; Influenza in Birds

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- 1 (Experimental): 100 subjects 45 mcg of influenza A/H5N1.
  Interventions: Biological: Influenza A/H5N1 Vaccine
- 2 (Placebo Comparator): 20 subjects saline placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Influenza A/H5N1 Vaccine — Monovalent inactivated subvirion influenza H5N1 vaccine (derived from A/Vietnam/1203/04). Packaged in single-dose vials of 90 mcg/mL (0.7 mL/vial). Dosage 45 mcg/0.5 mL administered intramuscularly.
  Arms: 1
Drug: Placebo — Normal saline administered intramuscularly.
  Arms: 2

SUMMARY:
The purposes of this study are: to make sure that there are no serious side effects of an experimental inactivated influenza A/H5N1 vaccine in children; and to see how the body's immune system reacts to the vaccine. To look at the side effects, researchers will follow children closely after vaccination. To look at immune system responses, researchers will test the children's blood before and a number of times after vaccination. Participants will include up to 130 healthy children ages 2-9 years. Participants will be assigned to receive 2, up to 3 doses of vaccine, or placebo (inactive substance). Subjects will receive at least 2 doses of vaccine approximately 28 days apart. If data shows an enhanced immune response from a third vaccination, children will be offered a third dose of the vaccine. Participants will be involved in study related procedures for up to 13 months, including up to 6 study visits, plus a number of telephone calls.

DETAILED DESCRIPTION:
The goals of this study are to assess the safety, reactogenicity, and immunogenicity of 45-microgram dosage level of monovalent subvirion influenza A/H5N1 virus vaccine administered by intramuscular (IM) route to healthy children. The primary goal of this study is to determine if this dosage level of H5N1 will result in an acceptable proportion of children achieving a potentially protective post vaccination antibody titer (provisionally assigned as a serum neutralizing titer of 1:40, based on studies conducted in Hong Kong during the 1997 H5N1 outbreak). Approximately 130 healthy children, aged 2 through 9 years, will be enrolled in this multicenter, randomized, double-blinded, placebo-controlled, clinical trial to receive at least 2 and up to 3 doses of an inactivated influenza A/H5N1 vaccine at a 45-microgram dose. One hundred subjects will be enrolled and randomly assigned into the influenza A/H5N1 vaccine dose group and 20 subjects into the placebo group (in 5:1 ratio). Subjects will be stratified into 2 age groups (2 to 5 years old and 6 to 9 years old). Vaccine or placebo will be administered into the deltoid. Subjects randomized to receive vaccine will receive 2 doses of the vaccine approximately 28 days apart. At approximately month 5, subjects' parent(s) or guardian(s) will be called to remind them of the 6-month follow-up visit. At the 6-month visit, subjects will be assessed for serious adverse events (SAEs) and the randomization assignment, ie, to vaccine or placebo, will be unmasked to the subject and parent(s) or guardian(s). Should data evaluating a third dose of the influenza A/H5N1 vaccine in adults show enhanced immunogenicity, parents or guardians of subjects who received vaccine will be offered a third dose, with an additional blood draw immediately prior to the third dose and 28 days and 6 months thereafter. The 6-month post-Dose 3 blood draw is optional. For subjects assigned to placebo, the parents or guardians will be offered the opportunity to enroll the subject into a separate open-label protocol if the 2 dose regimen administered to the vaccine recipients is found to be safe and immunogenic. The primary endpoints of the study include: adverse event (AE) and SAE information (solicited in-clinic and via memory aids, concomitant medications, and periodic targeted physical assessments, as indicated); proportion of subjects achieving a serum neutralizing antibody titer of 1:40 against the influenza A/H5N1 virus 28 days after receipt of second dose of vaccine (approximately Day 56); and geometric mean titer (GMT) and the frequency of 4-fold or greater increases in hemagglutination inhibition and neutralizing antibody titers 28 days after receipt of second dose of vaccine (approximately Day 56). The secondary endpoints of the study include: proportion of subjects achieving a serum neutralizing antibody titer of 1:40 against the influenza A/H5N1 virus 1 and 6 months after receipt of first and third doses (if third dose will be administered [see study design]) of vaccine; GMT and the frequency of 4-fold or greater increases in serum hemagglutination inhibition antibody titer 1 and 6 months after receipt of first and third (if third dose will be administered [see study design]) doses of vaccine; and development of serum antibody responses against antigenically drifted variants of influenza H5N1 virus. This study is linked to protocol 06-0072.

ELIGIBILITY:
Inclusion Criteria:

* The subject must be male or female, aged 2 through 9 years at enrollment.
* The subject must be in good health (and not on any chronic medications), as determined by medical history and a history-directed targeted physical examination.
* Parents or guardians must be able to understand and comply with planned study procedures and be available for all study visits.
* Parents or guardians must provide written consent prior to initiation of any study procedures, and subject may provide written assent as appropriate.

Exclusion Criteria:

* The subject must not have a known allergy to eggs or other components of the vaccine or sensitivity or allergy to latex.
* The subject must not have a history of asthma or recurrent wheezing.
* The subject must not be undergoing immunosuppression as a result of an underlying illness or treatment.
* The subject must not have an active neoplastic disease or a history of any hematologic malignancy.
* The subject must not be using oral or parenteral steroids, inhaled steroids, or other immunosuppressive or cytotoxic drugs. Note: Subjects on nasal or topical steroids will be allowed to enroll in this study.
* The subject must not have a history of receiving immunoglobulin or other blood product within the 3 months prior to enrollment in this study.
* The subject must not have received any other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrollment in this study.
* The subject must not have an acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe or would interfere with the evaluation of responses (these conditions include, but are not limited to, known chronic liver disease, significant renal disease, unstable or progressive neurological disorders, diabetes mellitus, and transplant recipients).
* The subject must not have a history of severe reactions following immunization with contemporary influenza virus vaccines.
* The subject must not have an acute illness, including an axillary temperature greater than 100 degrees F, within 3 days prior to vaccination.
* The subject must not have received an experimental vaccine or medication within one month prior to enrollment in this study, or expect to receive an experimental vaccine, medication, or blood product during the 13-month study period.
* The subject must not have any condition that would, in the opinion of the investigator, place them at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.
* History of Guillain-Barré syndrome.
* The subject must not be participating concurrently in another clinical trial (either in active phase or in follow-up phase).

Ages: 2 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 157 (Actual)
Dates: Start 2006-01; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Adverse event (AE) and serious adverse event (SAE) information (solicited in clinic and via memory aids, concomitant medications, and periodic targeted physical assessments.) | Solicited AEs-reactogenicity following each vaccination. Unsolicited AEs-SAEs occurring during the length of the study, and nonserious events occurring 28 days after receipt of the 2nd (from enrollment) or 3rd dose of vaccine.
Proportion of subjects achieving a serum neutralizing antibody titer of 1:40 against the influenza A/H5N1 virus. | 28 days after receipt of the 2nd dose of vaccine (Day 56).
Geometric mean titer and the frequency of 4-fold or greater increases in hemagglutination inhibition and neutralizing antibody titers. | 28 days after receipt of the 2nd dose of vaccine (Day 56).

SECONDARY OUTCOMES:
Proportion of subjects achieving a serum neutralizing antibody titer of 1:40 against the influenza A/H5N1 virus. | 1 and 6 months after receipt of first and third doses (if third dose will be administered [see study design]) of vaccine.
Geometric mean titer and the frequency of 4-fold or greater increases in serum hemagglutination inhibition antibody titer. | 1 and 6 months after receipt of first and third (if third dose will be administered [see study design]) doses of vaccine.
Development of serum antibody responses against antigenically drifted variants of influenza H5N1 virus. | Blood samples for serum assays will be collected at day 0, approximately 1 month after each immunization, and approximately 6 months after the first immunization and third immunization (if provided).

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - UCLA Center For Vaccine Research, Torrance, California
  - University of Maryland Baltimore, Baltimore, Maryland
  - Saint Louis University, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio